CLINICAL TRIAL: NCT03057925
Title: Ultrasound-guided Percutaneous Microwave Ablation for Benign Thyroid Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenjun Wu (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Wenjun Wu, associate chief physician, First Affiliated Hospital of Wenzhou Medical University
Organization: First Affiliated Hospital of Wenzhou Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wwju127
Record Dates: First submitted 2017-02-12; First posted 2017-02-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Thyroid Nodule
Keywords: thyroid nodule; microwave ablation
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): MWA Percutaneous Microwave Ablation intervention procedure: Ultrasound-guided Percutaneous Microwave Ablation
  Interventions: Device: Microwave Ablation
- Group B (No Intervention): untreated no treatment; regular ultrasonic image follow-up

INTERVENTIONS:
Device: Microwave Ablation — Ultrasound-guided Percutaneous Microwave Ablation
  Other Names: Ultrasound-guided Percutaneous Microwave Ablation
  Arms: Group A

SUMMARY:
Percutaneous microwave ablation(MWA) was reported as an effective modality for the management of thyroid nodules(TNs). This study aims to validate MWA as a feasible approach for patients with TNs for whom surgery is contraindicated or refused. Two groups of subjects with TNs(one group to treat with MWA and the other group to receive regular ultrasonic follow-up without any treatment) will be evaluated in term of TN volume, ultrasonic image and clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* benign thyroid nodules(TYP 2)
* solid or predominantly solid(colloid component<30%)large (>3.0ml) thyroid nodules
* refusal and/or inefficacy of surgery

Exclusion Criteria:

* pregnancy
* malignant or suspicious thyroid nodules

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the thyroid nodule volume assessed by ultrasonography after treatment vs simple clinical observation | From time to treatment until 12 months. Time point evaluations at 1,3,6,12 months
  Change of the thyroid nodule volume assessed by using ultrasonography, the volume reduction ratio(VRR) was calculated by the equation: VRR%=[(initial volume-final volume)*100]/initial volume

SECONDARY OUTCOMES:
Improved score on TN-related symptoms | From time to treatment until 12 months. Time point evaluations at 1,3,6,12 months
  Evaluation of TN-related neck symptoms scored separately as follow:0(absent),1(moderate),2(severe). The sum of the individual scores generates a final score(SYS score) ranging from 0 to 6
Improved cosmetic grading score | From time to treatment until 12 months. Time point evaluations at 1,3,6,12 months
  Cosmetic problem evaluated by grading score(1,no palpable mass;2, no cosmetic problem but palpable mass; 3, a cosmetic problem on swallowing only; and 4, a readily detected cosmetic problem

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Chen, Principal Investigator — Thyroid Center of The First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu W, Gong X, Zhou Q, Chen X, Chen X. Ultrasound-Guided Percutaneous Microwave Ablation for Solid Benign Thyroid Nodules: Comparison of MWA versus Control Group. Int J Endocrinol. 2017;2017:9724090. doi: 10.1155/2017/9724090. Epub 2017 Nov 23. PMID 29333159